CLINICAL TRIAL: NCT02472730
Title: Cap Assisted Colonoscopy Enhances Quality Based Competency in Colonoscopy Among Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Alliance for Academic Internal Medicine (Other)
Responsible Party: Principal Investigator, Kalpesh Patel, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-36849
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Endoscopy, Gastrointestinal
Keywords: Colonoscopy; Training Techniques; Endoscopy, Gastrointestinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cap Assisted Colonoscopy (Experimental): The distal attachment cap is affixed to the colonoscope before every colonoscopy in this arm.
  Interventions: Device: Distal Attachment Cap
- Standard Colonoscopy (No Intervention): Standard colonoscopy without the distal attachment cap is performed in this arm.

INTERVENTIONS:
Device: Distal Attachment Cap — Colonoscopies are performed under the supervision of board certified attending gastroenterologists experienced in colonoscopy. Attending physicians will provide assistance at their discretion or at the request of the trainee. All close examinations for polyps will be carried out on withdrawal of the colonoscope.
  Other Names: US Endoscopy Distal Attachment Cap
  Arms: Cap Assisted Colonoscopy

SUMMARY:
The purpose of this study is to identify if performing diagnostic colonoscopy with a small plastic cap attached to the camera will improve performance of colonoscopies by physician trainees.

DETAILED DESCRIPTION:
Training novice endoscopists to perform effective diagnostic colonoscopy is a central objective of Gastroenterology fellowship. Though there is no universal definition of competency, it is traditionally assessed with a combination of objective measures such as volume of procedures and subjective factors such as formal evaluations. As quality measures such as cecal intubation time, cecal intubation rate, and adenoma detection rate gain in importance in clinical practice, they should be increasingly incorporated as objectives into more formalized and objective training methodologies.

Indeed, though 140 colonoscopies have been suggested as a rough volume threshold needed for trainees to gain competence, evidence suggests that the number may actually be much higher when taking various objective quality measures into account.

Recent attention has turned to various measures to improve trainee performance such as computer simulation and magnetic endoscopy imaging. Along these lines, simple, effective, and economical measures are needed to improve trainee performance.

Cap assisted colonoscopy (CAC) is performed with the aid of a transparent inert cap attached to the distal end of the colonoscope. CAC allows close examination of mucosa proximal to flexures and haustral folds and prevents "red out" when closely approximated against mucosa, aiding in luminal orientation and examination. CAC has been shown to improve cecal intubation time, polyp detection rate, and adenoma detection rate in the hands of experienced practitioners. A handful of studies have also indicated that these benefits also extend to trainees, while another prospective study showed no improvement in cecal intubation rate.

The investigators hypothesize that cap assisted colonoscopy will result in significantly improved cecal intubation rate and time, as well as adenoma detection rate, among trainees when compared with standard non cap assisted colonoscopy in a large academic Gastroenterology training program in the United States.

The study is a prospective randomized trial of colonoscopies performed at Harris Health System Ben Taub Hospital by all novice endoscopy trainees from July 2015 until enrollment is complete. Novice endoscopy trainees are defined as endoscopists with less than 10 colonoscopies performed by July 2015. All colonoscopies included will be performed by the novice endoscopist under direct supervision of a board certified attending gastroenterologist.

Each colonoscopy fulfilling the inclusion criteria will be randomized with equal probability to a cap assisted colonoscopy (CAC) group or a control standard colonoscopy (SC) group.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing colonoscopy by a novice endoscopist

Exclusion Criteria:

* Age less than 18 years or greater than 90 years.
* Pregnancy.
* Prior surgical resection of colon or rectum.
* Known obstructing colorectal tumors.
* Severe hematochezia.
* Diverticulitis within 1 month of procedure.
* Clinical or radiological evidence of colonic obstruction or megacolon within 1 month of procedure.
* Referral for endoscopic mucosal resection.
* Unsedated colonoscopies.
* Colonoscopies abandoned due to inadequate bowel prep or colonoscopies with Boston bowel prep score < 3.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalpesh Patel, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

REFERENCES:
- [Background] ASGE Training Committee; Adler DG, Bakis G, Coyle WJ, DeGregorio B, Dua KS, Lee LS, McHenry L Jr, Pais SA, Rajan E, Sedlack RE, Shami VM, Faulx AL. Principles of training in GI endoscopy. Gastrointest Endosc. 2012 Feb;75(2):231-5. doi: 10.1016/j.gie.2011.09.008. Epub 2011 Dec 7. No abstract available. PMID 22154419
- [Background] Rex DK, Petrini JL, Baron TH, Chak A, Cohen J, Deal SE, Hoffman B, Jacobson BC, Mergener K, Petersen BT, Safdi MA, Faigel DO, Pike IM. Quality indicators for colonoscopy. Gastrointest Endosc. 2006 Apr;63(4 Suppl):S16-28. doi: 10.1016/j.gie.2006.02.021. No abstract available. PMID 16564908
- [Background] Vennes JA, Ament M, Boyce HW Jr, Cotton PB, Jensen DM, Ravich WJ, Sugawa C, Wu WC, Sanowski RA, Ament M, et al. Principles of training in gastrointestinal endoscopy. American Society for Gastrointestinal Endoscopy. Standards of Training Committees. 1989-1990. Gastrointest Endosc. 1992 Nov-Dec;38(6):743-6. No abstract available. PMID 1473697
- [Background] Sedlack RE. Training to competency in colonoscopy: assessing and defining competency standards. Gastrointest Endosc. 2011 Aug;74(2):355-366.e1-2. doi: 10.1016/j.gie.2011.02.019. Epub 2011 Apr 23. PMID 21514931
- [Background] Ward ST, Mohammed MA, Walt R, Valori R, Ismail T, Dunckley P. An analysis of the learning curve to achieve competency at colonoscopy using the JETS database. Gut. 2014 Nov;63(11):1746-54. doi: 10.1136/gutjnl-2013-305973. Epub 2014 Jan 27. PMID 24470280
- [Background] Gomez V, Wallace MB. Training and teaching innovations in colonoscopy. Gastroenterol Clin North Am. 2013 Sep;42(3):659-70. doi: 10.1016/j.gtc.2013.05.001. PMID 23931865
- [Background] Ng SC, Tsoi KK, Hirai HW, Lee YT, Wu JC, Sung JJ, Chan FK, Lau JY. The efficacy of cap-assisted colonoscopy in polyp detection and cecal intubation: a meta-analysis of randomized controlled trials. Am J Gastroenterol. 2012 Aug;107(8):1165-73. doi: 10.1038/ajg.2012.135. Epub 2012 Jun 5. PMID 22664471
- [Background] Rastogi A, Bansal A, Rao DS, Gupta N, Wani SB, Shipe T, Gaddam S, Singh V, Sharma P. Higher adenoma detection rates with cap-assisted colonoscopy: a randomised controlled trial. Gut. 2012 Mar;61(3):402-8. doi: 10.1136/gutjnl-2011-300187. Epub 2011 Oct 13. PMID 21997547
- [Background] Park SM, Lee SH, Shin KY, Heo J, Sung SH, Park SH, Choi SY, Lee DW, Park HG, Lee HS, Jeon SW, Kim SK, Jung MK. The cap-assisted technique enhances colonoscopy training: prospective randomized study of six trainees. Surg Endosc. 2012 Oct;26(10):2939-43. doi: 10.1007/s00464-012-2288-2. Epub 2012 Apr 27. PMID 22538693
- [Background] Manta R, Mangiavillano B, Fedeli P, Viaggi P, Castellani D, Conigliaro R, Masci E, Bassotti G. Hood colonoscopy in trainees: a useful adjunct to improve the performance. Dig Dis Sci. 2012 Oct;57(10):2675-9. doi: 10.1007/s10620-012-2213-5. Epub 2012 May 13. PMID 22581341
- [Background] Dai J, Feng N, Lu H, Li XB, Yang CH, Ge ZZ. Transparent cap improves patients' tolerance of colonoscopy and shortens examination time by inexperienced endoscopists. J Dig Dis. 2010 Dec;11(6):364-8. doi: 10.1111/j.1751-2980.2010.00460.x. PMID 21091899
- [Background] Prachayakul V, Aswakul P, Limsrivilai J, Anuchapreeda S, Bhanthumkomol P, Sripongpun P, Prangboonyarat T, Kachintorn U. Benefit of "transparent soft-short-hood on the scope" for colonoscopy among experienced gastroenterologists and gastroenterologist trainee: a randomized, controlled trial. Surg Endosc. 2012 Apr;26(4):1041-6. doi: 10.1007/s00464-011-1992-7. Epub 2011 Nov 1. PMID 22042588
- [Background] Kondo S, Yamaji Y, Watabe H, Yamada A, Sugimoto T, Ohta M, Ogura K, Okamoto M, Yoshida H, Kawabe T, Omata M. A randomized controlled trial evaluating the usefulness of a transparent hood attached to the tip of the colonoscope. Am J Gastroenterol. 2007 Jan;102(1):75-81. doi: 10.1111/j.1572-0241.2006.00897.x. Epub 2006 Nov 13. PMID 17100978
- [Background] Tee HP, Corte C, Al-Ghamdi H, Prakoso E, Darke J, Chettiar R, Rahman W, Davison S, Griffin SP, Selby WS, Kaffes AJ. Prospective randomized controlled trial evaluating cap-assisted colonoscopy vs standard colonoscopy. World J Gastroenterol. 2010 Aug 21;16(31):3905-10. doi: 10.3748/wjg.v16.i31.3905. PMID 20712051
- [Derived] Tang Z, Zhang DS, Thrift AP, Patel KK. Impact of cap-assisted colonoscopy on the learning curve and quality in colonoscopy: a randomized controlled trial. Gastrointest Endosc. 2018 Mar;87(3):723-732.e3. doi: 10.1016/j.gie.2017.06.011. Epub 2017 Jun 23. PMID 28648577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cap Assisted Colonoscopy | Standard Colonoscopy
Started | 110 | 109
Completed | 101 | 102
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cap Assisted Colonoscopy | Standard Colonoscopy | Total
Number analyzed (Participants) | 110 | 109 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 92 | 182
  >=65 years | 20 | 017 | 37
Age, Continuous [Median (Standard Deviation); unit: years] | 55.6 (8.84) | 55.8 (9.39) | 55.7 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Drop out due to clinical reasons
  Participants
    Female | 78 | 69 | 147
    Male | 32 | 40 | 72
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 110 | 109 | 219

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Successfully Reached the Cecum Within 30 Minutes of Insertion
Description: Proportion of all colonoscopies in which the trainee successfully reached the cecum within 30 minutes of insertion without the help of the attending physician.
Time Frame: Each outcome measured during a complete colonoscopy. All colonoscopies performed during the initial 3 months of a 12 month training program
Measure: Count of Participants; unit: Participants
Arm/Group | Cap Assisted Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 101 | 102
Participants | 80 | 67

2. Secondary Outcome: Mean Time From the Moment of Colonoscope Insertion Until the Appendiceal Orifice or Ileocecal Valve is Identified
Description: Time from the moment of colonoscope insertion until the appendiceal orifice or ileocecal valve is identified
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Cap Assisted Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 101 | 102
minutes | 13.7 [12.3 to 15.2] | 16.5 [14.7 to 18.2]

3. Secondary Outcome: Number of Colonoscopies During Which at Least One Adenoma Was Identified
Description: Proportion of colonoscopies that identify at least one adenoma
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cap Assisted Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 101 | 102
Participants | 38 | 44

4. Secondary Outcome: Number of Colonoscopies During Which at Least One Polyp Was Identified
Description: Proportion of colonoscopies that identify at least one polyp
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cap Assisted Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 101 | 102
Participants | 54 | 55

ADVERSE EVENTS:
Arm/Group | Cap Assisted Colonoscopy | Standard Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/102
Other Adverse Events (participants affected / at risk) | 0/101 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes